CLINICAL TRIAL: NCT05901246
Title: Anti-eryptotic Effect of Regular Intake of a Food Supplement with Plants Sterols in Subjects with Hypercholesterolemia Treated with Statins
Brief Title: Anti-eryptotic Effect of a Food Supplement with Plants Sterols in Hypercholesterolemia Treated with Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other); University of Bologna (Other)
Responsible Party: Principal Investigator, Amparo Alegria, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIONUTEST_2023/069; PID2019-104167RB-I00 (Other Grant/Funding Number: MCIN/AEI/10.13039/501100011033)
Record Dates: First submitted 2023-05-08; First posted 2023-06-13 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases; Hypercholesterolemia; Atherosclerosis
Keywords: Cholesterol; Plant Sterols; Eryptosis; Cholesterol oxidation products
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PS-containing dietary supplement (Experimental): Sachet containing a powdered ingredient source of microencapsulated free plant sterols (2,25 g ingredient/day)
  Interventions: Dietary Supplement: PS-containing dietary supplement
- Placebo (Placebo Comparator): Sachet containing the excipients of the ingredient (2,25 g placebo/day)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: PS-containing dietary supplement — Sachet containing a powdered ingredient source of microencapsulated free plant sterols (2,25 g ingredient/day)
  Arms: PS-containing dietary supplement
Other: Placebo — Sachet containing the excipients of the ingredient (2,25 g placebo/day)
  Arms: Placebo

SUMMARY:
Potential anti-eryptotic effect of a regular intake of a plant sterol (PS)-containing food supplement, in moderate hypercholesterolemic patients treated with the PS-containing food supplement or placebo supplement.

DETAILED DESCRIPTION:
Oxidative damage has been related to the externalization of phosphatidylserine in erythrocytes, an event associated with eryptosis (programmed death of erythrocytes). In addition, an increase in eryptosis has been observed in patients with hypercholesterolaemia. PS-enriched food supplements could be a nutritional strategy to improve risk factors in patients with moderate hypercholesterolemia treated with statins, constituting a synergistic treatment with these drugs. The present study aims to evaluate the eryptotic process (externalization of phosphatidylserine) after regular intake of a food supplement containing PS (2g/day) in patients with moderate hypercholesterolemia treated with statins. This is a case-control study with 32 cases (intake or a PS-containing food supplement) and 16 controls (placebo intake based on the excipient), with an intervention period of 6 weeks. The evaluation of eryptosis is carried out by determining the externalization of phosphatidylserine, the size of the erythrocytes and an ex vivo assay of adhesion of eryptotic erythrocytes to the vascular endothelium. In addition, the redox state (GSH), the in vivo oxidation of cholesterol (COPs), and biochemical and hematological parameters are evaluated. All parameters are evaluated at the beginning (week 0) and at the end of the intervention period (week 6).

ELIGIBILITY:
Inclusion Criteria:

* Participants with hypercholesterolemia (LDL cholesterol ≥ 160mg/dl at the time of diagnosis), receiving treatment with moderate intensity statins (atorvastatin 10-20 mg or simvastatin 20-40 mg or rosuvastatin 5-10 mg)
* No previous episodes of cardiovascular disease
* Absence of other analytical abnormalities or previous illnesses

Exclusion Criteria:

* Diabetes mellitus
* Participants in secondary prevention
* Treatment with lipid-lowering drugs other than atorvastatin, simvastatin or rosuvastatin
* Liver disease
* Renal failure
* Uncontrolled hypothyroidism
* Smokers
* Participants consuming foods enriched with PS or food supplements that contain PS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Changes in the externalization of phosphatidylserine | 0 and 6 weeks
  The externalization of phosphatidylserine, assessed by flow cytometry (Kit Annexin V) with repeated measures (at the beginning and at the end of the intervention)
Changes in the adhesion to the endothelium by eryptotic erythrocytes | 0 and 6 weeks
  The adhesion to the endothelium by eryptotic erythrocytes, assessed with parallel-plate flow chamber technique in human umbilical vein endothelial cells (HUVECs) with repeated measures (at the beginning and at the end of the intervention)

SECONDARY OUTCOMES:
Changes in cell size ('forward scatter') | 0 and 6 weeks
  Cell size, assessed by flow cytometry with repeated measures (at the beginning and at the end of the intervention)
Changes in reduced glutathione cellular levels (GSH) | 0 and 6 weeks
  GSH, assessed by flow cytometry (Green CMFDA), with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic levels of cholesterol oxidation products (COPs) | 0 and 6 weeks
  COPs levels, assessed by gas chromatography-mass spectometry, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic glucose | 0 and 6 weeks
  Glucose, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic total cholesterol | 0 and 6 weeks
  Total cholesterol, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic HDL-c | 0 and 6 weeks
  HDL-c, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic LDL-c | 0 and 6 weeks
  LDL-c, calculated by the Friedewald's formula, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic triglycerides | 0 and 6 weeks
  Triglycerides, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic Apo A | 0 and 6 weeks
  Apo A, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic Apo B | 0 and 6 weeks
  Apo B, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic High-sensitivity C-reactive protein (hsCRP) | 0 and 6 weeks
  hs CRP, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic insulin | 0 and 6 weeks
  Insulin, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Changes in plasmatic Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 0 and 6 weeks
  HOMA-IR, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of the intervention)
Evaluation of the mediterranean diet adherence to measure quality of life | 0 weeks
  Mediterranean diet adherence screener (MEDAS) is used, consisting in 14 questions (each one 0 or 1 point, final score between 0 and 14). Results are ranged between 0-7 points (low adherence), 7-10 (moderate adherence), and 10-14 (high adherence). This is only evaluated at the beginning of the intervention.
Evaluation of the physical activity to measure quality of life | 0 weeks
  International physical activity questionaire-short form (IPAC-SF) is used, consisting in 7 questions. Intensity, frequency and duration of the exercise are evaluated through metabolic equivalent of task (METs). This allows to differentiate 3 levels of physical activity:
  Low: Not enough activity to achieve the next level
  Moderate: 3 or more days of vigorous physical activity for at least 20 minutes per day, 5 or more days of moderate physical activity and/or walking at least 30 minutes per day, or 5 or more days of any combination of walking, moderate or vigorous physical activity achieving at least a total of 600 METs
  High: Vigorous physical activity at least 3 days per week achieving a total of at least 1500 METs, or 7 days of any combination of walking, with moderate and/or vigorous physical activity, achieving a total of at least 3000 METs
  This is only evaluated at the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Asunción Alegría Torán, Professor, Principal Investigator — University of Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cilla A, Lopez-Garcia G, Collado-Diaz V, Amparo Blanch-Ruiz M, Garcia-Llatas G, Barbera R, Martinez-Cuesta MA, Real JT, Alvarez A, Martinez-Hervas S. Hypercholesterolemic patients have higher eryptosis and erythrocyte adhesion to human endothelium independently of statin therapy. Int J Clin Pract. 2021 Nov;75(11):e14771. doi: 10.1111/ijcp.14771. Epub 2021 Sep 7. PMID 34473881
- [Background] Restivo I, Attanzio A, Tesoriere L, Allegra M, Garcia-Llatas G, Cilla A. Anti-Eryptotic Activity of Food-Derived Phytochemicals and Natural Compounds. Int J Mol Sci. 2022 Mar 11;23(6):3019. doi: 10.3390/ijms23063019. PMID 35328440